CLINICAL TRIAL: NCT06970561
Title: Analysis of Factors Associated With Postoperative Recurrence of Intraductal Papilloma of the Breast Treated With Ultrasound-guided Vacuum-assisted Rotary Excision
Brief Title: Analysis of Recurrence of Intraductal Papilloma Treated With Vacuum-assisted Rotary Excision
Acronym: IDP
Status: Completed | Type: Observational
Sponsor: Wuhan Children's Hospital (Other)
Responsible Party: Principal Investigator, Gang Hu, Attending physician，Thyroid and breast surgery, Wuhan Children's Hospital
Other Study IDs: 2020091
Record Dates: First submitted 2025-05-04; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Surgery; Benign Breast Tumors
Keywords: intraductal papilloma of the breast; treatment; vacuum-assisted rotational excision therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- recurrent: Patients who relapsed after receiving ultrasound-guided vacuum-assisted rotary excision
  Interventions: Procedure: enlarged resection
- non-recurrent: Patients who did not relapsed after receiving ultrasound-guided vacuum-assisted rotary excision

INTERVENTIONS:
Procedure: enlarged resection — patients underwent secondary enlarged resection within 1 month after the diagnosis of IDP combined with ADH,
  Other Names: secondary enlarged resection
  Groups: recurrent

SUMMARY:
To study the postoperative recurrence of intraductal papillomas (IDP) treated with ultrasound-guided vacuum-assisted excision (VAE), and to investigate the effect of different lesion characteristics on recurrence.

DETAILED DESCRIPTION:
106 patients with IDP with or without atypical ductal hyperplasia (ADH) treated with ultrasound-guided VAE at Zhongnan Hospital of Wuhan University from January 2020 to August 2024 were selected for the study, and the postoperative conditions of the patients were sorted out and followed up to analyze the characteristics of the lesions and to determine the relevant factors that affected the postoperative recurrence.

ELIGIBILITY:
Inclusion Criteria:

* IDP was diagnosed pathologically after VAE treatment
* the tumor was a solitary lesion with the margin >1cm from the nipple and the longest diameter of the tumor <3cm
* it was not associated with other breast diseases

Exclusion Criteria:

* previous ductal breast surgery
* abnormal coagulation function or taking anticoagulant drugs .recent or current use of hormonal or psychotropic drugs.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IDP patients who underwent ultrasound-guided VAE treatment from January 2020 to August 2024 in Zhongnan Hospital of Wu han University.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
recurrence | The cut-off date for follow-up was September 2024
  Recurrence was defined as the appearance of a lesion within 2-3 cm of the original surgical area with corresponding clinical manifestations, such as nipple discharge and imaging support, which was later pathologically confirmed as IDP

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: starting 6 months after publication
Access Criteria: The IPD can be shared for the summary report of test results,the reanalysis of test data and enables the combination of test data with other data for new research.